CLINICAL TRIAL: NCT02702934
Title: Metabolic Effects of High-amylose Wheat-based Rusks in Healthy Subjects. A Pilot Study.
Brief Title: Metabolic Effects of High-amylose Wheat-based Rusks.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, Professor, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 233/14
Record Dates: First submitted 2016-03-02; First posted 2016-03-09 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2016-03

CONDITIONS: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-amylose rusks (Experimental): Test meal with 100g of carbohydrates coming from high-amylose rusks
  Interventions: Other: Test meal
- Control rusks (Active Comparator): Test meal with 100g of carbohydrates coming from regular rusks used as control
  Interventions: Other: Test meal

INTERVENTIONS:
Other: Test meal — Participants received in random order a test meal (900Kcal, 100g carbohydrates) containing rusks prepared with amylose-rich wheat flour or conventional flour. Blood samples were collected at fasting and every 30 minutes over 4 hours. Breath hydrogen was evaluated as a marker of intestinal fermentation. Participants underwent Visual Analogue Scale to assess subjective appetite sensations.
  Other Names: Acute test meal

SUMMARY:
Amylose-amylopectin ratio may influence the rate of starch digestion. This randomized controlled study evaluated the postprandial metabolic effects of amylose-rich- wheat- based rusks in overweight subjects.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese;
* 30-60 years.

Exclusion Criteria:

* age <30 and >60 years;
* fasting triglycerides ≥400 mg/dl;
* fasting cholesterol >270 mg/dl;
* cardiovascular events (myocardial infarction or stroke) during the 6 months prior to the study;
* established diabetes mellitus or any chronic disease;
* renal and liver failure (creatinine >1.7 mg/dl and transaminases >2 times than normal values, respectively);
* anaemia (Hb <12 g /dl);
* any chronic disease.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Blood glucose | 4 hours
  Incremental area under the curve

SECONDARY OUTCOMES:
Blood insulin | 4 hours
  Incremental area under the curve
Intestinal fermentation | 4 hours
  Incremental area under the curve
Blood triglycerides | 4 hours
  Incremental area under the curve

CONTACTS AND LOCATIONS:
Overall Officials: Angela Rivellese, Professor, Principal Investigator — Federico II University
Locations (1):
- Department of Clinical Medicine and Surgery, Naples, Italy

IPD SHARING:
Plan to Share IPD: No